CLINICAL TRIAL: NCT05540405
Title: A Randomized, Double-blind, Controlled, Parallel-arm Trial to Assess the Effects of a Bitter Melon Product at Two Doses vs. Control on Indicators of Cardiometabolic Health in Men and Women With Prediabetes
Brief Title: Effects of Bitter Melon on Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Greenyn Biotechnology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MB-2202
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose bitter melon (Experimental): Subject will receive 1 Insumate bitter melon capsule/d (300 mg) and 1 placebo capsule/d (300 mg)
  Interventions: Dietary Supplement: Low-dose bitter melon
- High-dose bitter melon (Experimental): Subject will receive 2 Insumate bitter melon capsules/d (300 mg each)
  Interventions: Dietary Supplement: High-dose bitter melon
- Placebo (Placebo Comparator): Subject will receive 2 placebo capsules/d (300 mg each)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Low-dose bitter melon — Subject will receive 1 Insumate bitter melon capsule/d (300 mg) and 1 placebo capsule/d (300 mg)
  Arms: Low-dose bitter melon
Dietary Supplement: High-dose bitter melon — Subject will receive 2 Insumate bitter melon capsules/d (300 mg each)
  Arms: High-dose bitter melon
Dietary Supplement: Placebo — Subject will receive 2 placebo capsules/d (300 mg each)
  Arms: Placebo

SUMMARY:
The objectives of this study are to assess the effects of a bitter melon product at two doses, compared to control, on indicators of cardiometabolic health among men and women with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 74 years of age, inclusive.
2. Subject has BMI 25.00 to 39.99 kg/m2, inclusive.
3. Subject has prediabetes defined as fasting capillary glucose 100 to 125 mg/dL, inclusive, and/or HbA1c 5.7% to 6.4%, inclusive, at screening.
4. Subject is judged by the Investigator to be in generally good health on the basis of medical history and screening measurements.
5. Subject is willing to abstain from consumption of bitter melon (other than the study products) throughout the study.
6. Subject is willing and able to undergo the scheduled study procedures.
7. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject has consumed a bitter melon food or product within 8 weeks prior to the screening visit (week -1) (washout permitted).
2. Subject has a laboratory test result of clinical significance based on the judgment of the Principal Investigator or qualified designee.
3. Subject has a clinically significant medical condition that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
4. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at screening.
5. Subject has a history of cancer in the prior 5 years, except non-melanoma skin cancer or carcinoma in situ of the cervix.
6. Subject has had a weight change of +/-4.5 kg (10 lbs) in the previous 3 months.
7. Subject has extreme dietary habits (e.g., Atkins, vegan, very low carbohydrate diet).
8. Subject has a history of bariatric surgery, is currently taking a weight loss drug, or is actively attempting to lose or gain body weight.
9. Subject has taken a proprotein convertase subtilisin kexin type 9 (PCSK9) inhibitor agent within 12 weeks prior to screening.
10. Subject has unstable use (defined as initiation or change in dose) of the following lipid-altering medications within 4 weeks prior to screening: bile acid sequestrants, fibrates, niacin (drug form), statins, ezetimibe, bempedoic acid, or omega-3-ethyl ester drugs.
11. Subject has taken any hypoglycemic medications within 4 weeks prior to screening including: insulin, sodium-glucose cotransporter-2 (SGLT2)-inhibitors, alpha-glucosidase inhibitors, biguanides, thiazolidinediones, dipeptidyl peptidase-4 (DPP-4) inhibitors, meglitinides, sulfonylureas, glucagon-like peptide-1 (GLP-1) receptor agonists, GLP-1/glucose-dependent insulinotropic polypeptide (GIP) modulators.
12. Subject has unstable use (defined as initiation or change in dose) of anti-hypertensive medications within 4 weeks prior to screening.
13. Subject has used systemic corticosteroids within 4 weeks prior to screening.
14. Subject has taken dietary supplements meant to regulate carbohydrate or lipid metabolism or body weight, within 4 weeks of screening, including, but not limited to, chromium picolinate, ginseng, starch blockers, omega-3 fatty acid supplements (e.g., flaxseed, fish or algal oils), red rice yeast supplements, garlic supplements, soy isoflavone supplements, niacin or its analogues at doses >400 mg/day, plant sterol or stanols, and/or irregular or inconsistent use of Metamucil® or other viscous fiber-containing supplements (consistent, daily use up to 1 teaspoon of a viscous-fiber supplement is acceptable).
15. Subject has signs or symptoms of an active infection of clinical significance or has taken antibiotics within 5 days prior to any visit (washout is permitted for re-scheduling of the clinic visit).
16. Subject has an allergy, sensitivity or intolerance to any components of the study products.
17. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
18. Subject has been exposed to any non-registered drug product within 30 days prior to screening.
19. Subject has a current or recent history (within 12 months prior to screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
20. Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | Baseline to 12 weeks
  Change in HbA1c

SECONDARY OUTCOMES:
Glycated hemoglobin (HbA1c) | Baseline to 6 weeks
  Change in HbA1c
Fasting glucose | Baseline up to 12 weeks
  Change in fasting glucose
Fasting insulin | Baseline up to 12 weeks
  Change in fasting insulin
Homeostasis model assessment of insulin sensitivity (HOMA%S) | Baseline up to 12 weeks
  Change in HOMA%S
Homeostasis model assessment of beta-cell function (HOMA%B) | Baseline up to 12 weeks
  Change in HOMA%B
Total cholesterol | Baseline up to 12 weeks
  Change in total cholesterol
Low-density lipoprotein cholesterol (LDL-C) | Baseline up to 12 weeks
  Change in LDL-C
High-density lipoprotein cholesterol (HDL-C) | Baseline up to 12 weeks
  Change in HDL-C
Non-HDL-C | Baseline up to 12 weeks
  Change in non-HDL-C
Fasting triglycerides | Baseline up to 12 weeks
  Change in triglycerides
Body fat | Baseline up to 12 weeks
  Change in body fat
Skeletal muscle mass | Baseline up to 12 weeks
  Change in skeletal muscle mass

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — MB Clinical Research & Consulting
Locations (3):
- United States (3):
  - Excellence Medical & Research, Miami Gardens, Florida
  - Health Awareness, Port Saint Lucie, Florida
  - Biofortis, Inc., Addison, Illinois

IPD SHARING:
Plan to Share IPD: No